CLINICAL TRIAL: NCT01517815
Title: Pharmacokinetic of Doripenem and Piperacillin/Tazobactam in More Than 120 kg Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8739
Record Dates: First submitted 2012-01-11; First posted 2012-01-25 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2013-11

CONDITIONS: Septic Shock
Keywords: Septic shock; overweight; critically ill; pharmacokinetic; doripenem; piperacillin-tazobactam
MeSH Terms: conditions — Shock, Septic; Overweight; Critical Illness | interventions — Doripenem; Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No overweight patient (Experimental): Patient with weight less than or equal to 120kg
  Interventions: Drug: Doripenem or Piperacillin/Tazobactam
- Overweight patients (Experimental): Patient with weight more than 120kg
  Interventions: Drug: Doripenem or Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Doripenem or Piperacillin/Tazobactam — This arm is composed of 26 no overweight patients, Antibiotic (Doripenem or Piperacillin/Tazobactam) is chosen by the intensivist in charge of the case:
  * in 13 no overweight patients, Pipéracilline/tazobactam will be administered in 4g IV (1h) and then 16g/24h IV continuously. Piperacillin/Tazobactam plasma dosage: after the first dose and then every 12h.
  * in 13 patients no overweight: doripénème will be administered in 1g/8h with a 4h IV infusion. Doripenem plasma dosage: after the first dose and then twice a day, at peak and residual value.
  Other Names: no overweight patients pharmacokinetics
  Arms: No overweight patient
Drug: Doripenem or Piperacillin/Tazobactam — This arm is composed of 26 overweight patients, Antibiotic (Doripenem or Piperacillin/Tazobactam) is chosen by the intensivist in charge of the case:
  * in 13 overweight patients, Pipéracilline/tazobactam will be administered in 4g IV (1h) and then 16g/24h IV continuously. Piperacillin/Tazobactam plasma dosage: after the first dose and then every 12h.
  * in 13 patients overweight: doripénème will be administered in 1g/8h with a 4h IV infusion. Doripenem plasma dosage: after the first dose and then twice a day, at peak and residual value.
  Other Names: overweight patients pharmacokinetics
  Arms: Overweight patients

SUMMARY:
Overweight patients are susceptible to develop acute complications when they are admitted in an Intensive Care Unit (ICU). Severe infection can be associated with cardiovascular failure ('shock") and is associated with 35-50% mortality. One of the key issue to cure infection is to administer antibiotics. However, under dosing antibiotic is one of the main reason that explain treatment failure. There are very few data concerning particularities of antibiotic dosing in critically ill, overweight, patients. The aim of the present study is to describe the pharmacokinetic of two main antibiotics (doripenem and piperacillin/Tazobactam) in both overweight and non overweight critically ill patients presenting a septic shock. The investigators hypothesis is that usual dose for those antibiotic may be accurate in non overweight patients but is not in overweight patients.

DETAILED DESCRIPTION:
N=52 patients divided in 4*13 patients (13 per antibiotic and per group, overweight or non overweight).

Overweight is defined by a weight over 120kg. Antibiotic chosen by the intensivist in charge of the case. Doripenem 1g/8h with a 4h IV infusion whatever the patient's weight. Piperacillin/Tazobactam 4g IV (1h) and then 16g/24h IV continuously whatever the patient's weight.

Piperacillin/Tazobactam plasma dosage: after the first dose and then every 12h. Doripenem plasma dosage: after the first dose and then twice a day, at peak and residual value.

Usual plasma and urine samples for urea, creatinine, electrolytes, platelets and bilirubin each 24h.

Microbiology: bacterial identification and MIC measurement with E-test

ELIGIBILITY:
Inclusion Criteria:

General:

* Patients in severe sepsis or septic shock defined by Bone criteria (proved or very suspected infection with organ impairment and/or need of vasopressive agent to keep a mean arterial pressure more than 65mmHg)
* Patient requiring a treatment by study's antibiotics
* Informed consent signed
* Patient must be affiliated or beneficiary of a social medical insurance
* Participation of patient to the trial must be noted in the medical file

Specific to overweight patients: Weight > 120kg

Specific to no overweight patients: Weight less than or equal to 120kg

Exclusion Criteria:

* Pregnant women
* Under age patient minor
* Patient protected by law
* Known allergy to study's antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time over MIC (calculated with the E-test) in overweight and non overweight critically ill patients | up to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Boris BJ JUNG, MD, Principal Investigator — Saint Eloi Hospital - Montpellier University Hospital
Locations (1):
- Saint Eloi Intensive Care Unit - Montpellier University Hospital, Montpellier, France